CLINICAL TRIAL: NCT06163118
Title: Validation of a Screening Tool for Swallowing Disorders for the Elderly
Acronym: DéGluT'G
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21_RIPH2-14
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-11

CONDITIONS: Swallowing Disorder; Dysphagia
Keywords: Swallowing Disorder; Dysphagia; Swallowing Disorder test; Bronchopneumonia; Geriatric short-stay unit
MeSH Terms: conditions — Deglutition Disorders; Bronchopneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient aged 75 or over hospitalized in the Geriatric Short-Stay Unit (Experimental): Two caregivers from the Geriatric Short-Stay Unit will successively administer the "Deglut'G" tool to each patient, blind to each other, and blind to the SLP and ENT doctor examination. All patients will have a SLP examination and an ENT doctor examination aimed at detecting swallowing disorders.
  Interventions: Diagnostic Test: Deglut'G test; Diagnostic Test: SLP swallowing test; Diagnostic Test: ENT doctor swallowing test

INTERVENTIONS:
Diagnostic Test: Deglut'G test — Two tests to assess swallowing disorders using the Deglut'G tool will be carried out by a nurse or a caregiver from the Geriatric Short-Stay Unit, at visit 1.
  The tests can be taken successively, or spaced apart by a time defined by the medical team, and will be taken blind to each other.
  The average test administration time will be measured during the study, but the test should not exceed 10 minutes depending on the patients.
  The Deglut'G tool consists of an initial administration of gelled water (1 to 3 teaspoons), to identify if a cough occurs. In the event of a cough, the oral treatment is stopped; if the cough is absent, a new step this time consists of the administration of water (1 to 3 sips). In case of cough, the food will be mixed, the liquids thickened, and the medicinal treatments crushed. If there is no cough, foods and liquids can be taken as normal.
Diagnostic Test: SLP swallowing test — At visit 1, 1 to 2 hours after the last Deglut'G test, a second swallowing test will be carried out by a SLP according to his skills and according to his usual practice, independently of the Deglut'G tool.
  This test should not exceed 20-30 minutes depending on the patient.
Diagnostic Test: ENT doctor swallowing test — At Visit 2 (day 7 +/- 3 days after the inclusion), still as part of the short-stay hospitalization, the patient will meet an ENT doctor who will carry out an examination aimed at detecting swallowing disorders, according to his usual practice, of independent of the Deglut'G tool.
  The examination should not exceed 20-30 minutes depending on the patient.

SUMMARY:
Swallowing disorder, or dysphagia, is a lack of protection of the airways during the passage of the food bolus towards the esophagus. Swallowing disorder is characterized by a feeling of discomfort when swallowing, difficult swallowing in elderly people or a blockage felt during the progression of food between the mouth and the stomach, sometimes with falsities. These disorders can be the cause of a loss of appetite and a reduction in food consumption in older people.

In the most serious cases, they can lead to aspiration, weakening the pulmonary passages and possibly leading to suffocation.

Swallowing disorders constitute an important public health problem due to their prevalence among the elderly. Many early readmissions could be avoided thanks to better quality of care in these patients.

In the elderly, the number of comorbidities and the multiplicity of medications and drug intake increase the incidence of swallowing disorders in this population. They constitute a common pathology, probably underestimated and underdiagnosed in the geriatric population.

Given the aging of the Martinique population, it is appropriate to offer an easy-to-use, quickly achievable tool for diagnostic purposes, making it possible to quickly identify potential swallowing disorders, and therefore to anticipate meal intake, and on the adaptation of the prescription to a medicinal alternative (before any food or medication taken during hospitalization).

In the Geriatric Short-Stay Unit of the Martinique University Hospital, a tool called "Deglut'G", was developed, and has been used since 2015, in order to allow caregivers a rapid, reliable and relevant assessment of swallowing disorders in the elderly, in order to guide care and medication alternatives.It now appears important to validate this tool, by comparing it with the results of examinations of swallowing disorders obtained from a speech-language pathologists (SLPs) and an ENT doctor.

ELIGIBILITY:
Inclusion Criteria:

* Person aged 75 or over hospitalized in the Geriatric Short-Stay Unit,
* Person having been informed of the research,
* Person having given free written and informed consent,
* Person affiliated to a social security scheme.

Exclusion Criteria:

* Person unable to take the tests,
* Person with an oral condition that hinders normal swallowing (stomatitis, gingivitis, etc.),
* Elderly person under legal protection, under guardianship or curatorship,
* Person who refused to participate in the study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Measure the concordance between the results of the SLP examination, and those obtained with the Deglut'G tool, for the detection of swallowing disorders. | 12 months
  Concordance between the results of the Deglut'G test and the SLP assessment.
  The evaluation of a swallowing disorder via the DegluT'G tool, by the geriatric short-stay unit caregivers, will be done as follows:
  * Presence of cough following administration of gelled water : suspicion of swallowing disorder
  * Presence of cough following administration of water : suspicion of swallowing disorder
  * Absence of cough following administration of water : no swallowing disorder
  This assessment will be compared to the SLP assessment, whatever the assessment method used.

SECONDARY OUTCOMES:
Measure the concordance between the results of the ENT doctor examination, and those obtained with the Deglut'G tool, for the detection of swallowing disorders | 12 months
  Concordance between the results of the Deglut'G test and the ENT doctor assessment.
  The evaluation of a swallowing disorder via the DegluT'G tool, by the geriatric short-stay unit caregivers, will be done as follows:
  * Presence of cough following administration of gelled water : suspicion of swallowing disorder
  * Presence of cough following administration of water : suspicion of swallowing disorder
  * Absence of cough following administration of water : no swallowing disorder
  This assessment will be compared to the ENT doctor assessment, whatever the assessment method used.
Measure the concordance of the measurements obtained with the Deglut'G tool between two caregivers, for the detection of swallowing disorders | 12 months
  Inter-rater reliability of Deglut'G screening
Estimate the average time it takes to use the Deglut'G tool | 12 months
  Time taken to take the Déglut'G tests (in minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Seendy Bartholet, PhD, Principal Investigator — University Hospital Center of Martinique
Locations (1):
- University Hospital Center of Martinique, Fort-de-France, France